CLINICAL TRIAL: NCT05679583
Title: Preoperative Stereotactic Body Radiation Therapy in Patients With Resectable Pancreatic Cancer: A Prospective Phase II Study
Brief Title: Preoperative Stereotactic Body Radiation Therapy in Patients With Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-1062
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative SBRT arm (Experimental): Patients with resectable pancreatic cancer will receive preoperative SBRT 2 to 4 weeks before surgery. And 4 weeks after surgery, adjuvant CTx will be administered for 6 months.
  Interventions: Radiation: Preoperative Stereotactic body radiation therapy (SBRT), Pancreatic resection, Adjuvant Chemotherapy

INTERVENTIONS:
Radiation: Preoperative Stereotactic body radiation therapy (SBRT), Pancreatic resection, Adjuvant Chemotherapy — 1. Preoperative Stereotactic body radiation therapy (SBRT) For the gross pancreatic cancer lesion, 30 Gy/5 fx will be prescribed considering respiratory movement. And 20 Gy/5 fx will be prescribed to the triangle operation area including the common hepatic artery, celiac artery, and portal vein.
  2. Pancreatic resection Surgical resection will be performed 2-4 weeks after the end of radiation therapy. The surgical method and resection range depend on the surgeon's judgment at the time of surgery.
  3. Adjuvant Chemotherapy Adjuvant chemotherapy will be given under the judgment of the oncologist from 4 weeks after surgical resection, considering the pathological findings (R0 or R1 resection status, etc.) and the patient's medical condition. Adjuvant chemotherapy includes gemcitabine alone, gemcitabine plus capecitabine combination therapy, and mFOLFIRINOX.

SUMMARY:
Pancreatic cancer is a cancer with a poor prognosis and a high mortality rate. The prognosis of surgically resectable pancreatic cancer is better than that of unresectable pancreatic cancer. But the prognosis is still poor enough to report a 2-year disease-free survival rate of 47.0% despite the application of standard treatment. Preoperative chemotherapy or radiotherapy for pancreatic cancer has been performed for a long time, especially for locally advanced pancreatic cancer. However, there are very few studies on the application of preoperative chemotherapy or radiotherapy for borderline resectable or resectable pancreatic cancer. The PREOPANC trial is a representative randomized study to investigate the effect of preoperative chemo/radiation therapy in borderline resectable or resectable pancreatic cancer. As a result, the overall survival, progression-free survival, local control, and distant control rates were significantly superior in preoperative therapy group. However, when only patients with resectable pancreatic cancer were analyzed separately, there was no significant difference in overall survival rate or complete resection rate. In 2020, retrospective propensity score matching analysis using the national cancer database revealed that the addition of preoperative stereotactic body radiation therapy (SBRT) showed a significant increase in overall survival rate rather than preoperative chemotherapy alone. In addition, SBRT also showed a significant increase in overall survival rather than conventional fractionated RT. In summary, the current standard treatment for resectable pancreatic cancer is surgical resection, but a higher survival rate can be expected when preoperative therapy is added. However, there is no study that focused on the role of preoperative SBRT. Therefore, this study aims to confirm the effectiveness of adding preoperative SBRT alone in resectable pancreatic cancer.

ELIGIBILITY:
Inclusion criteria:

1. Histologically diagnosed adenocarcinoma of the pancreas
2. Resectable pancreatic cancer at the time of diagnosis

   * Resectable pancreatic cancer refers to cases in which all of the following conditions are met:

     1. If the tumor does not reach the superior mesenteric vein or portal vein, or even if it does, it reaches within 180°
     2. If the tumor does not reach the superior mesenteric artery, celiac artery, or common hepatic artery
     3. In the absence of distant metastases 3) Patients aged 20 years or older at the time of diagnosis 4) General performance status is 0-2 based on the Eastern Cooperative Oncology Group (ECOG) standard 5) Patients who voluntarily decided to participate in this clinical study and signed the written informed consent

Exclusion criteria:

1. If there is a history of radiation exposure to the abdomen
2. Pancreatic cancer that cannot be resected
3. When accompanied by distant metastasis
4. Patients who are currently judged to be difficult to undergo surgery based on general performance status, bone marrow, and kidney function tests
5. Patients with active or uncontrolled infection
6. Patients with uncontrolled heart disease
7. Pregnant or lactating women
8. Patients with a history of malignant tumor excluding skin epithelial carcinoma, except for malignant melanoma, stage 0 cervical cancer, and early thyroid cancer
9. Patients who have been treated for malignant tumors and have been cured for more than 5 years can participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
R0 rate | 2 weeks after the surgical resection
  R0 resection is defined as the resection margin more than 1 mm away from the tumor on histological findings after pancreatic cancer surgery. The R0 rate refers to the proportion of patients showing R0 resection, based on all patients.

SECONDARY OUTCOMES:
Disease-free survival | Patient follow-up will be performed 3 months after the surgery and then at 6-month intervals thereafter. Follow-up will be conducted for a total of 2 years.
  Disease-free survival It is based on the time from the date when pancreatic cancer was first diagnosed histologically to the time when recurrence was confirmed on clinical or radiological examination or when the subject died.
Local control rate | Patient follow-up will be performed 3 months after the surgery and then at 6-month intervals thereafter. Follow-up will be conducted for a total of 2 years.
  Local control rate It is based on the time from the date when pancreatic cancer was first diagnosed histologically to the time when local recurrence was confirmed on clinical and radiological examination.
Overall survival rate | Patient follow-up will be performed 3 months after the surgery and then at 6-month intervals thereafter. Follow-up will be conducted for a total of 2 years.
  Overall survival rate It is based on the date from the date of the first histological diagnosis of pancreatic cancer to the date of death of the subject or the date of the last follow-up.
Treatment related acute/chronic toxicity (based on CTCAE ver 5.0) | Patient follow-up will be performed 3 months after the surgery and then at 6-month intervals thereafter. Follow-up will be conducted for a total of 2 years.
  Treatment related acute/chronic toxicity (based on CTCAE ver 5.0) During treatment, immediately after the end of treatment, 3 months after treatment, and at 6-month intervals thereafter, CTCAE 5.0 is measured.
Quality of life (based on EORTC QLQ-C30) | Patient follow-up will be performed 3 months after the surgery and then at 6-month intervals thereafter. Follow-up will be conducted for a total of 2 years.
  Quality of life (based on EORTC QLQ-C30) Before the start of treatment, immediately after completion, 3 months after treatment, and every 6 months until 2 years thereafter.
Quality of life (based on FACT-Hep) | Patient follow-up will be performed 3 months after the surgery and then at 6-month intervals thereafter. Follow-up will be conducted for a total of 2 years.
  Quality of life (based on FACT-Hep) Before the start of treatment, immediately after completion, 3 months after treatment, and every 6 months until 2 years thereafter.
Tumor recurrence | Patient follow-up will be performed 3 months after the surgery and then at 6-month intervals thereafter. Follow-up will be conducted for a total of 2 years.
  Tumor recurrence Imaging tests and tumor marker tests are performed every 3-6 months after treatment to determine the presence or absence of tumor recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Ik Jae Lee, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No